CLINICAL TRIAL: NCT04103606
Title: A Mobile-App Training to Reduce Body Image Disorder Symptoms and Associated Psychological Features in Female University Students: a Randomized Controlled Pilot Study with Crossover Design
Brief Title: A Mobile-App Training to Reduce Body Image Disorder Symptoms and Associated Features in Female University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Silvia Cerea, Postdoctoral Research Fellow, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2936
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2022-12

CONDITIONS: Body Image Disorder; Body Dysmorphic Disorders; Eating Disorders
MeSH Terms: conditions — Body Dysmorphic Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate-use App group (iApp group) (Experimental): Participants in the iApp group start using the app immediately (Time 0; T0) for 16 consecutive days (until Time 1; T1).
  Interventions: Device: GGBI: Positive Body Image (Mobile App)
- delayed-use App group (dApp) (Active Comparator): Participants in the dApp group start using the app at Time 1 (T1; 16 days after the iApp group) and use the app for the following 16 days (Time 2; T2).
  Interventions: Device: GGBI: Positive Body Image (Mobile App)

INTERVENTIONS:
Device: GGBI: Positive Body Image (Mobile App) — Brief, game-like, training exercise for challenging body image disorder symptoms and associated psychological features

SUMMARY:
Body dissatisfaction represents a prevalent condition in young women, and it is associated with low self-esteem, depression, and symptoms of Body Dysmorphic Disorder (BDD) and Eating Disorders (EDs). The aim of the trial is to test the effect of a mobile health application called "GGBI: Positive Body Image" in reducing body dissatisfaction, body dysmorphic disorder/eating disorder symptoms, and associated psychological features in female university students considered at high-risk of developing Body Image Disorders (BIDs).

Hypothesis: Participants using "GGBI: Positive Body Image" immediately following baseline assessment (Time 0; T0) (immediate-use App group: iApp) would exhibit greater reduction in body dissatisfaction, body dysmorphic disorder/eating disorder symptoms, and associated psychological features than participants who did not use "GGBI: Positive Body Image" in this phase of the study (delayed-use App group: dApp). Following crossover (Time 1; T1), the investigators expect that participants gains in the iApp group would be maintained at follow-up (Time 2; T2).

ELIGIBILITY:
Inclusion Criteria:

* Presence of Body Image Disorder symptoms

Exclusion Criteria:

* Presence of a full-blown Body Image Disorder
* Presence of a psychotic/schizophrenic disorder
* Current treatment for a Body Image Disorder

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change of body dissatisfaction and body dysmorphic disorder symptoms | 16 days
  Assessed with the Questionario sul Dismorfmismo Corporo (Questionnaire about Body Dysmorphic Disorder; QDC; Cerea et al., 2017), a self-report questionnaire assessing body dissatisfaction and body dysmorphic disorder symptoms made up of 40 items. Items are rated on a 7-point Likert scale (from 1 = strongly disagree to 7 = strongly agree; score range: 40-280), with higher scores indicating extreme body dissatisfaction and body dysmorphic disorder symptoms. Individuals who score above the cut-off of the questionnaire (QDC total score = 130) should be referred for further assessment because they might present extreme body dissatisfaction/body dysmorphic disorder symptoms or may be at risk of developing body dysmorphic disorder
Change of eating attitudes and behaviors | 16 days
  Eating Disorder Inventory-3 (EDI-3; Garner, 2004; Italian version by Giannini et al., 2008): a self-report questionnaire assessing eating disorders core features made up of 91 items on a 6-point Likert scale (from always to never), with higher scores indicating higher eating disorder symptoms. It contains three primary subscales: Drive for Thinness (score range = 0-28; higher scores indicating higher drive for thinness), Bulimia (score range = 0-32; higher scores indicating higher bulimic symptoms), and Body Dissatisfaction (score range = 0-40; higher scores indicating higher body dissatisfaction). These subscales compose the Eating Disorder Risk Composite (EDRC) score. The other nine additional scales are Low Self-Esteem, Personal Alienation, Interpersonal Insecurity, Interpersonal Alienation, Interoceptive Deficits, Emotional Dysregulation, Perfectionism, Asceticism, and Maturity Fears.

SECONDARY OUTCOMES:
Change of self-esteem | 16 days
  Assessed with the Rosenberg Self Esteem Scale (RSES; Rosenberg, 1965; Italian version by Prezza, Trombaccia, and Armento, 1997), a self-report questionnaire assessing self-esteem. The Rosenberg Self Esteem Scale is made up of 10 items rated on a 4-point Likert scale (from 1 = "strongly disagree" to 4 = "strongly agree" ), with higher scores indicating higher self-esteem
Change in social anxiety symptoms | 16 days
  Assessed with the Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998; Italian version by Sica, Musoni, Bisi, Lolli, & Sighinolfi, 2007), a self-report questionnaire assessing social anxiety symptoms. The Social Interaction Anxiety Scale made up of 19 items on a 5-point Likert scale (from 0 = "not at all characteristic of true of me" to 4 = "extremely characteristic of true of me"; score range: 0-76); higher scores indicate higher levels of social interaction anxiety symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padua, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Yes